CLINICAL TRIAL: NCT00636038
Title: Bioavailability of Yellow Maize Carotenoids in Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Nutricia Research Fundation (Other); National University of Science and Technology, Zimbabwe (Other)
Responsible Party: Guangwen Tang, Tufts University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2007-E6
Record Dates: First submitted 2008-03-07; First posted 2008-03-14 (Estimated); Last update posted 2008-03-14 (Estimated); Status verified 2008-03

CONDITIONS: Vitamin A Status
Keywords: beta-carotene; yellow maize; vitamin A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: corn beta-carotene — yellow corn beta-carotene in a 1 mg level to be taken as corn porridge in one meal by volunteers
  Other Names: staple food beta-carotene

SUMMARY:
The study hypothesis is that high ß-C yellow maize can provide vitamin A efficiently.

- list item one ß-C in yellow maize

The study will use stable isotope labeled high ß-C yellow maize and vitamin A in a well-nourished population by utilizing stable isotope dilution techniques. In this project, deuterium labeled vitamin A that is derived from the labeled ß-C yellow maize will be traced after being eaten by a human subject. Eight men (> 40 years and < 70 y) who are healthy, non-smoking,body weight within 20% of standard weight for height (Metropolitan) and not having taken vitamin A or ß-C supplements within the last month will be recruited as volunteers. This study will last for 50 days during which at day 1, cooked labeled yellow maize paste (porridge) equal to a total of ~ 2 bowls cooked yellow maize (from 100 - 200 g dry weight) containing ~ 1 mg ß-C will be taken by each volunteer. On day 8, a labeled vitamin A (1 mg of 13C retinyl acetate) in oil dose will be used in evaluation of liver storage of vitamin A. Forty six blood samples (460 cc) will be taken during the study which will be analyzed for serum carotenoids and retinoids using HPLC and mass spectrometry techniques.

The serum concentration and isotope ratio of ß-C and retinol will be determined. Serum enrichment curve following each oral dose will be studied. The area under the curve (AUC) of retinol-d4 and labeled retinol from the reference dose in serum samples will be determined and compared. The equivalence of a high ß-C corn meal to vitamin A will be calculated based on the isotope reference method to determine the efficiency of corn ß-C to provide vitamin A.

DETAILED DESCRIPTION:
- list item one ß-C in yellow maize

Pro-vitamin A carotenoids in plants are a major and safe vitamin A source for a vast population in the world. Even though, ß-carotene (ß-C) in vegetables has been considered as a safe vitamin A source, it is essential to determine the efficiency of provitamin A carotenoids in plant conversion to vitamin A. However, the bioavailability of vitamin A and carotenoids from food matrices has not been well studied due to the unavailability of isotopically labeled foods that can be fed to humans.

The main objective of this study is to investigate the bioavailability of ß-C in yellow maize and its bioconversion to retinol stored in the liver using stable isotope labeled high ß-C yellow maize and vitamin A in a well-nourished population by utilizing stable isotope dilution techniques. In this project, the deuterium labeled vitamin A that is derived from the labeled ß-C yellow maize will be traced after being eaten by a human subject. This will allow for quantitative determination of the vitamin A equivalence of high ß-C plant foods.

Eight men (> 40 years and < 70 y) who are healthy, non-smoking adults must have their body weight within 20% of standard weight for height (Metropolitan) and not having taken vitamin A or ß-C supplements within the last month will be recruited as volunteers.

This is a 50 day study during which dose 1, cooked labeled yellow maize paste (porridge) equal to a total of ~ 2 bowls cooked yellow maize (from 100 - 200 g dry weight) containing ~ 1 mg ß-C will be taken by each volunteer. On day 8, dose 2 will be used in evaluation of liver storage of vitamin A using 1 mg of 13C retinyl acetate. One blood sample (20 cc) will be drawn during the screening process. Forty six blood samples (460 cc) will be taken during the study which will be analyzed for serum carotenoids and retinoids using HPLC and mass spectrometry techniques. The serum concentration and isotope ratio of ß-C and retinol will be determined. Serum enrichment curve following each oral dose will be studied. The area under the curve (AUC) of retinol-d4 and labeled retinol from the reference dose in serum samples will be determined and compared. The equivalence of a high ß-C plant food supplement to a vitamin A dose will be calculated based on the isotope reference method.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects

Exclusion Criteria:

* GI track problems

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Bioavailability of corn beta-carotene and its equivalency to provide vitamin A | one year

CONTACTS AND LOCATIONS:
Locations (1):
- National University of Science and Technology, Bulawayo, Zimbabwe

REFERENCES:
- [Derived] Muzhingi T, Gadaga TH, Siwela AH, Grusak MA, Russell RM, Tang G. Yellow maize with high beta-carotene is an effective source of vitamin A in healthy Zimbabwean men. Am J Clin Nutr. 2011 Aug;94(2):510-9. doi: 10.3945/ajcn.110.006486. Epub 2011 Jun 29. PMID 21715509